CLINICAL TRIAL: NCT03240952
Title: Establishing Reference Range for Community-dwelling Elderly Nutrition
Brief Title: The Nutritional Health for the Elderly Reference Centre Study (NHERC Study)
Acronym: NHERC
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: Changi General Hospital (Other); SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Other Study IDs: BL35 (Part 1)
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elderly are at greater risk of dietary insufficiency due to age-related increases in nutrient requirements concomitant with a reduction in energy requirements, decreases in appetite and energy intake. Currently there is a gap in knowledge of the factors that are associated with malnutrition in the elderly in Singapore. In addition, there is no "reference" database on anthropometric measurements and biochemical indices for elderly with a range of nutrition status in Singapore. Thus, the objectives of this cross-sectional study are to examine factors influencing nutritional status and to determine the reference values for anthropometric and biochemical measurements related to nutritional status for community-dwelling elderly in Singapore.

DETAILED DESCRIPTION:
This is a cross-sectional study. Measurements will be taken at baseline for elderly with normal nutrition (n = 400) and elderly who are at risk of under nutrition (n = 800).. These measurements will be used to examine factors influencing nutritional status and to create a "reference" database for anthropometric and biochemical measurements related to nutritional status for use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged ≥65 years.
2. Community-dweller, i.e. not staying in a residential intermediate and long-term care (ILTC) service institution.
3. Participant is being discharged home directly (applicable for hospital cohort).
4. Participant is community ambulant with or without aid.
5. Participant does not have any chronic disease(s) or has stable chronic disease(s) including hypertension, chronic obstructive pulmonary disease, and cardiovascular disease in the opinion of the Study Physician, at study entry.
6. Participant has voluntarily signed and dated an informed consent form (ICF), approved by an Institutional Review Board (IRB) and provided authorization prior to any participation in the study.
7. Participants will be able to communicate and follow instructions.
8. Participant is able to consume food and beverages orally.

Exclusion Criteria:

1. Participant has been diagnosed with dementia according to medical records.
2. Participant has been diagnosed with type 1 or type 2 diabetes according to medical records. (Note: This includes participant with controlled diabetes.)
3. Participant has any active infectious disease (such as tuberculosis, Hepatitis B or C, HIV infection) according to medical records.
4. Participant has been diagnosed with severe gastrointestinal disorders including celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis according to medical records.
5. Participant has been diagnosed with end stage organ or pre-terminal diseases or acute myocardial infarction within the last 30 days from the screening according to medical records.
6. Participant has malignancy according to medical records.
7. Participant has any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.
8. Participant is taking part in another study that has not been approved as a concomitant study by the study team.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This cross-sectional study will include 400 elderly with normal nutrition (MUST score: 0) and 800 elderly who are at risk of undernutrition (MUST score ≥ 1). Community-dwelling elderly recently discharged from the hospital as well as those who recently visited polyclinics in Singapore will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
MUST | Baseline
  Malnutrition risk using Malnutrition Universal Screening Tool

SECONDARY OUTCOMES:
Body weight, fat mass, fat free mass | Baseline
  Body weight, fat mass, fat free mass in kilograms will be measured using Tanita MC-780
Pre-albumin | Baseline
  Pre-albumin in mg/dL will be measured using Cobas
Albumin and total protein | Baseline
  Albumin and total protein in g/L will be measured using Cobas

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ling Tey, Ph.D., Study Chair — Abbott Nutrition Research & Development; Samuel TH Chew, MB.BCh.BAO, Principal Investigator — Changi General Hospital
Locations (4):
- Singapore (4):
  - Marine Parade Polyclinic, Singapore
  - Bedok Polyclinic, Singapore
  - Tampines Polyclinic, Singapore
  - Changi General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong RHS, Chow WL, Cheong M, Lim GH, Xie W, Baggs G, Huynh DTT, Oh HC, How CH, Tan NC, Tey SL, Chew STH. Associations between socio-demographics, nutrition knowledge, nutrition competencies and attitudes in community-dwelling healthy older adults in Singapore: findings from the SHIELD study. J Health Popul Nutr. 2021 Dec 11;40(1):52. doi: 10.1186/s41043-021-00277-4. PMID 34895351